CLINICAL TRIAL: NCT06082349
Title: Effectiveness and Cost-effectiveness of Lymphaticovenous Anastomosis for Cancer Patients Who Suffer From Chronic Peripheral Lymphedema: a Randomized Controlled Trial
Brief Title: The N-LVA Study: RCT Comparing LVA vs. Sham Surgery in Cancer-related Lymphedema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Radboud University Medical Center (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL84169.068.23; 2021038374 (Other Grant/Funding Number: ZonMw/Zorginstituut Nederland); METC23-023 (Other: Medical Ethical Committee azM/UM)
Record Dates: First submitted 2023-10-03; First posted 2023-10-13 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Lymphedema, Secondary; Lymphedema of Upper Limb; Lymphedema, Lower Limb; Lymphedema Arm; Lymphedema of Leg
Keywords: Lymphaticovenous anastomosis; Sham surgery; Microsurgery; LVA
MeSH Terms: conditions — Lymphedema; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Multicenter, double-blind, randomized sham-controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The researcher, research nurse and patients will be blinded. The blinded researcher and research nurse will perform the measurements during follow-up, as well as the assessment of the outcomes. Due to the nature of the study, the surgeon performing both procedures cannot be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lymphaticovenous anastomosis (LVA) (Experimental): Patients in this group will undergo lymphaticovenous anastomosis at one or more locations on the affected limb, and the procedure will be performed under local anesthesia. During the operation, patients will be blinded using a noise-canceling headphone and blindfolds. Incisions will be made at the sites where lymphatic vessels are obstructed, ensuring no harm to the viable part of the lymphatic system. The locations will be determined prior to the surgery using ICG lymphography. The LVA(s) will be made in the subdermal plane with the aid of a surgical microscope. Generally, 1 to 4 LVAs are made. The LVA(s) is made using a surgical microscope and the operation will take approximately 60 to 90 minutes.
  Interventions: Procedure: Lymphaticovenous anastomosis
- Sham surgery (Sham Comparator): Patients in this group will undergo sham surgery at one location on the affected limb, and the procedure will be performed under local anesthesia. During the operation, patients will be blinded using a noise-canceling headphone and blindfolds. The locations for LVA surgery will be determined prior to the surgery using ICG lymphography. However, the incision for the sham procedure will be made 2 centimeters medial or lateral to the predetermined site. This is done in order to avoid damage to the lymph vessels as to allow for future LVA surgery. After the incision, no LVA is made. Rather than performing the actual operation, the plastic surgeon will simulate the procedure by applying pressure in the surgical area. To mimic the approximate duration of a regular LVA procedure, the sham operation will take approximately 60 to 90 minutes.
  Interventions: Procedure: Sham surgery

INTERVENTIONS:
Procedure: Lymphaticovenous anastomosis — Lymphaticovenous anastomosis (LVA) involves connecting a lymphatic vessel to an adjacent vein of similar size, thereby facilitating the outflow of lymphatic fluid in patients suffering from secondary lymphedema
  Other Names: LVA; Lymphaticovenular anastomosis; Lymphovenous bypass; Lymphatic-venous shunt
  Arms: Lymphaticovenous anastomosis (LVA)
Procedure: Sham surgery — Sham surgery involves the process of surgery, including local anesthesia and incisions, but no LVA is made.
  Other Names: Placebo surgery; Simulated surgery; Surgical placebo
  Arms: Sham surgery

SUMMARY:
The goal of this randomized controlled trial is to compare the effectiveness and cost-effectiveness of lymphaticovenous anastomosis (LVA) with sham surgery for patients suffering from unilateral cancer-related lymphedema in either the upper or lower extremity. It aims to answer whether LVA is more effective than sham surgery in terms of improvement in Lymph-ICF score.

A total of 110 participants will be allocated randomly into two groups at a 1:1 ratio. The first group will receive lymphaticovenous anastomosis (LVA), while the second group will undergo sham surgery.

DETAILED DESCRIPTION:
One of the most debilitating side effects of cancer treatment is cancer-related lymphedema (CRL), with an overall incidence of 15.5%. To date, there is no definite cure for lymphedema. Conservative therapy, namely complex decongestive therapy is the golden standard for the treatment. Lymphaticovenous anastomosis (LVA) might be a promising treatment modality for patients with CRL, but available studies are small and the quality is lacking. No large-scale prospective or randomized studies have been published on the efficacy of LVA.

The main objective of this randomized controlled trial is to assess whether LVA is more effective than sham surgery in terms of improvement in Lymph-ICF score, volume reduction, reduction of complex decongestive therapy, and cost-effectiveness.

The study will take place in three centers in the Netherlands: Maastricht University Medical Center, Radboud University Medical Center, and Erasmus University Medical Center.

The patients will be randomly distributed into two groups: the LVA group or the Sham group. Both procedures are performed under local anesthesia. Patients in both groups are subject to minor surgical complications (wound infection, bleeding, wound dehiscence). Special care will be taken to prevent damage to lymphatic vessels in the Sham group, to allow a future LVA operation once the study ends. The follow-up moments will be at 3, 6, 12, 18, and 24 months. Additionally, a subset of patients will partake in an annual extended follow-up, ongoing until the start of the analysis. Each follow-up moment will last 45 minutes in total. The patient also receives two digital questionnaires at each follow-up moment.

ELIGIBILITY:
Inclusion Criteria:

* Treated for cancer and underwent treatment of either axillary or inguinal lymph nodes or radiotherapy;
* Early stage lymphedema (ISL I-II) in the upper or lower extremity, and diagnosed by lymphoscintigraphy for the lower extremity;
* Unilateral lymphedema;
* Viable lymphatic vessels as determined by indocyanine green (ICG)Lymphography (stage II-III);
* Refractory lymphedema that underwent at least three months of conservative treatment;
* Informed consent.

Exclusion Criteria:

* History of lymphatic reconstruction in the past 10 years;
* Late-stage lymphedema of the extremity (ISL classification ≥ II lymphedema) with evident fat deposition and/or fibrosis;
* Patients with active distant metastases, treated with palliative intent;
* Patients with the active treatment of primary cancer, i.e. surgery, radiotherapy, and/or chemotherapy. Note: patients receiving adjuvant targeted and/or endocrine treatment are eligible;
* Edema due to venous insufficiency, evaluated by venous duplex ultrasound of the deep and superficial venous system;
* Active infection in the lymphedematous extremity;
* Bilateral lymphedema;
* Lymphedema present in genital or breast area only;
* Primary lymphedema;
* Non-viable lymphatic system as determined by ICG Lymphography (stages IV and V).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Lymph-ICF Score at 12 and 24 months | Baseline, 3, 6, 12, 18 and 24 months post-operatively and afterwards annually during the extended follow-up, lasting up to the start of the first analysis (maximally 3 years extra or 3 additional visits).
  The Dutch version of the 'Lymphedema Functioning, Disability, and Health" (Lymph-ICF) questionnaire is used. There are two versions of the Lymph-ICF; one for the upper extremity and one for the lower extremity. The questionnaires assess the impairments in function, activity limitations, and participation restrictions of patients with lymphedema. It is a validated, disease-specific questionnaire, consisting of items across 5 domains. Each item is scored on a VAS, ranging from 0 to 100.

SECONDARY OUTCOMES:
Change from baseline in excess limb volume | Baseline, 3, 6, 12, 18 and 24 months post-operatively and afterwards annually during the extended follow-up, lasting up to the start of the first analysis (maximally 3 years extra or 3 additional visits).
  The excess limb volume will be measured with BioImpedance Spectroscopy (BIS). With a bioimpedance device, the volume of the extremities can be measured together with the fluid in different compartments of the extremities.
Change from baseline in extremity circumference measured by the Upper and Lower Extremity Lymphedema (UEL and LEL) indices | Baseline, 3, 6, 12, 18 and 24 months post-operatively and afterwards annually during the extended follow-up, lasting up to the start of the first analysis (maximally 3 years extra or 3 additional visits).
  The extremity circumference will be measured using measuring tape according to the fixed measuring points of the UEL- and LEL-indices. The UEL- and LEL-indices are corrected for BMI.
Change from baseline in the use of conservative treatment | Baseline, 3, 6, 12, 18 and 24 months post-operatively and afterwards annually during the extended follow-up, lasting up to the start of the first analysis (maximally 3 years extra or 3 additional visits).
  Discontinuation of conservative treatment, being complex decongestive therapy, will be assessed with a patient diary to record the frequency of treatments received (i.e. skin therapy visits, number of compression garments, etc.).
Postoperative complications | Baseline, 3, 6, 12, 18 and 24 months post-operatively and afterwards annually during the extended follow-up, lasting up to the start of the first analysis (maximally 3 years extra or 3 additional visits).
  All postoperative complications for both treatment groups will be recorded to monitor safety. SAEs will be directly reported to the sponsor.
Patency of the LVA | 12 and 24 months post-operatively and afterwards annually during the extended follow-up, lasting up to the start of the first analysis (maximally 3 years extra or 3 additional visits).
  The patency of the LVAs will be measured with ICG lymphography
Patient costs, QALYs, and incremental cost-effectiveness | Baseline, 3, 6, 12, 18 and 24 months post-operatively and afterwards annually during the extended follow-up, lasting up to the start of the first analysis (maximally 3 years extra or 3 additional visits).
  Patients costs are registered by the patient in the patient diary. The QALY will be calculated using the EQ-5D-5L questionnaire. The EQ-5D is a questionnaire responsive to changes in health in cancer-patients after the conclusion of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shan Shan Qiu Shao, MSc, PhD, Principal Investigator — Maastricht University Medical Center; Stefan Hummelink, MSc, PhD, Study Chair — Radboud University Medical Center; Dalibor Vasilic, MSc, PhD, Study Chair — Erasmus Medical Center
Locations (3):
- Netherlands (3):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Maastricht University Medical Center, Maastricht, Limburg
  - Erasmus University Medical Center, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: Yes
The results will be published under an Open Access license, making them accessible to everyone at all times. Requests for sharing individual participant data (IPD) will be evaluated on a case-by-case basis, assessing them for suitable research purposes following the trial's completion.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available upon request after the completion of the trial and publication of primary manuscripts. Individual participant data will be stored for a period of 15 years.
Access Criteria: Request for data sharing of individual participant data (IPD) will be assessed individually by the principal investigator, considering them for appropriate research purposes after the completion of the trial.

REFERENCES:
- [Background] Kleeven A, Jonis YMJ, Tielemans H, van Kuijk S, Kimman M, van der Hulst R, Vasilic D, Hummelink S, Qiu SS. The N-LVA Study: effectiveness and cost-effectiveness of lymphaticovenous anastomosis (LVA) for patients with cancer who suffer from chronic peripheral lymphoedema - study protocol of a multicentre, randomised sham-controlled trial. BMJ Open. 2024 Apr 15;14(4):e086226. doi: 10.1136/bmjopen-2024-086226. PMID 38626967
- See also: Study website — https://nlvastudy.com/